CLINICAL TRIAL: NCT02168829
Title: The Optimal Anticoagulation for Enhanced Risk Patients Post-Catheter Ablation for Atrial Fibrillation Trial
Brief Title: Optimal Anticoagulation for Higher Risk Patients Post-Catheter Ablation for Atrial Fibrillation Trial
Acronym: OCEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Bayer (Industry); Biotronik Canada Inc (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 327494
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: AF ablation; Anticoagulation AF ablation; Stroke prevention
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Active Comparator): Rivaroxaban 15 mg daily
  Interventions: Drug: Rivaroxaban
- Acetylsalicylic acid (ASA) (Active Comparator): ASA 75-160 mg daily (if intolerant to ASA, no antiplatelet therapy will be prescribed)
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Rivaroxaban
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Acetylsalicylic acid
  Other Names: Aspirin; ASA
  Arms: Acetylsalicylic acid (ASA)

SUMMARY:
This trial is comparing medical approaches for stroke prevention in people who have atrial fibrillation (AF) and have undergone a successful procedure called ablation to eliminate or substantially reduce the arrhythmia. AF is normally associated with an increased risk of stroke which in many patients can be prevented with appropriate blood thinner therapy. This trial will compare a strategy of oral anticoagulant therapy after successful ablation to therapy with an aspirin per day.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized trial to investigate whether a strategy of ongoing, long-term oral anticoagulation with rivaroxaban 15 mg daily is superior to a strategy of antiplatelet therapy, ASA 75-160 mg, alone in preventing cerebral embolic events in moderately high risk patients following successful catheter ablation for atrial fibrillation..

At least one year post-successful catheter ablation for AF or left atrial flutter/tachycardia without evidence of any clinically apparent arrhythmia recurrence based on at least one 24 hour Holter and ECG within 6 months after the last ablation procedure and at least one 24 hour Holter and ECG between 6 and 12 months post-ablation or beyond. Patient must have no atrial fibrillation, atrial flutter or atrial tachycardia > 30 seconds detected on a minimum 48 hour Holter monitor within two months prior to enrollment.

Patients will be randomized in a 1:1 fashion to ASA 75-160 mg daily or rivaroxaban 15 mg daily. Patients will be seen at 6 months, one year and every year thereafter for a minimum of 3 years. Blood chemistry tests, ECG, holters and patient quality of life questionnaires will be done annually.

Cerebral MRI scanning at baseline and at three years will be done for assessment of silent cerebral infarction. MRI imaging will be performed using a specific protocol.

A pre-specified subset of patients will undergo insertion of a implantable loop recorder (ILR) capable of automated AF detection.

ELIGIBILITY:
Inclusion Criteria

1. Patient must be at least one year post-successful catheter ablation(s) for atrial fibrillation without evidence of any clinically apparent arrhythmia recurrence defined as all of the following: No AF/AT/AFL on at least 24 hour Holter and an ECG (or equivalent) from 2-6 months after the last ablation, AND no AF/AT/AFL on at least 24 hour Holter and an ECG any time after 6 months after the last ablation AND no AF/AT/AFL on at least 24 hour Holter and ECG 2 months before enrolment in the study. The Holter/ECG within 2 months of enrolment may also serve as the Holter performed 6 months or later after the last ablation - see section 2.3.1 for details.
2. Patient must have a CHA2DS2-VASc risk score of 1 or more. Patients in whom female sex or vascular disease are their sole risk factor may not be enrolled.
3. Patient must be >18 years of age.
4. Patient must have non-valvular AF.

Exclusion Criteria

1. Patient does not meet all of the above listed inclusion criteria.
2. Patient is unable or unwilling to provide informed consent.
3. Patient is included in another randomized clinical trial or a clinical trial requiring an insurance.
4. Patient has been on an investigational drug within 30 days of enrolment.
5. Patient has been on strong CYP3A inducers (such as rifampicin, phenytoin, phenobarbital, or carbamazepine) or strong CYP3A inhibitors (such as ketoconazole or protease inhibitors) within 4 days of enrolment.
6. Patient has creatinine clearance < 30 mL/min.
7. Patient has bleeding contra-indication to oral anticoagulation (such as bleeding diathesis, hemorrhagic disorder, significant gastrointestinal bleeding within 6 months, intracranial/intraocular/ atraumatic bleeding history, fibrinolysis within 48 hours of enrollment).
8. Patient has other contraindication to oral anticoagulation or treatment with antiplatelet agent (such as allergy).
9. Patient has a contraindication to magnetic resonance imaging (MRI) or is unlikely to tolerate due to severe claustrophobia.
10. Patients with a contraindication to implantation of an implantable loop recorder if the patient opts for a loop recorder as part of the study (such as limited immunocompetence or a wound healing disorder).
11. Patient has valvular atrial fibrillation [reference AHA guidelines].
12. Patient has a non-arrhythmic condition necessitating long-term oral anticoagulation.
13. Patient had a severe, disabling stroke within one year prior to enrollment or any stroke within 14 days of enrollment.
14. Patient with special risk factors for stroke unrelated to AF, specifically known thrombophilia/ hypercoagulability, uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg within 4 days of enrollment), untreated familial hyperlipidemia, known vascular anomaly (intracranial aneurysm/ arteriovenous malformation or chronic vascular dissection), or known severe carotid disease.
15. Pregnancy or breastfeeding.
16. Women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception throughout the study.
17. Patients who are > 85 years of age.
18. Patients who are critically ill or who have a life expectancy <3 years.
19. Patients for whom the investigator believes that the trial is not in the interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Composite of stroke, systemic embolism and covert embolic stroke as detected by cerebral MRI | 3 years
  Composite of stroke, systemic embolism and covert embolic stroke as detected by cerebral MRI. A patient will be considered to have a covert stroke if one or more lesions > 15 mm has been detected between the baseline, and final (3 year) MRI on T2 weighted and/or FLAIR imaging protocols.

SECONDARY OUTCOMES:
Clinical, overt stroke | Up to 3 years
  Clinical, Overt stroke
Incidence of one or more covert MRI stroke(s) >15 mm | Up to 3 years
  Incidence of one or more covert MRI stroke(s) >15 mm
Composite of all major and minor bleeding | Up to 3 years
  Composite of all major and minor bleeding
Major bleeding only | Up to 3 years
  Major bleeding only
Minor bleeding only | Up to 3 years
  Minor bleeding only
Intracranial hemorrhage | Up to 3 years
  Intracranial hemorrhage (clinical and covert on MRI alone)
Transient ischemic attack | Up to 3 years
  Transient ischemic attack defined as presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting <24 hours
All-cause mortality | Up to 3 years
  All-cause mortality
Net clinical benefit based on reduction in stroke/TIA rate compared to major bleeding events. | Up to 3 years
  Net clinical benefit based on reduction in stroke/TIA rate compared to major bleeding events.
Occurrence of non-primary endpoint MRI changes from baseline to final scan | 3 years
  Occurrence of non-primary endpoint MRI changes from baseline to final scan including: quantification of cerebral atrophy, quantification of cerebral white matter changes, number of all new MRI lesions > 3mm, >5 mm, > 15 mm, and > 20 mm, and number of lesions detected exclusively on DW-MRI
Neuropsychological testing | 3 years
  Neuropsychological testing - performed at baseline and repeated at 3 years.
Health economics | 3 years
  Cost utilization and cost effectiveness analysis
Quality of life Assessment | Quality of Life is measured at Baseline and 36 months
  Quality of life Assessment measured with the Quality of life scale, EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Southlake Regional Health Centre; David H Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (55):
- Australia (5):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Melbourne, Melbourne, Victoria
  - Melbourne Health, Melbourne, Victoria
  - Heart Rhythm Clinic, Nedlands, Western Australia
- Belgium (16):
  - Algemeen Stedelijk Ziekenhuis - campus Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - Arlon - Clinique du Sud-Luxembourg, Arlon
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint-Jan (Brugge), Bruges
  - Europa Ziekenhuizen - ST-ELISABETH, Brussels
  - Sint-Jean - Kliniek Sint-Jan (Brussels), Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - Middelares Gent - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Ziekenhuis Oost-Limburg , campus St Jan, Lanaken
  - Universitair Ziekenhuis Leuven, campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - AZ Delta campus Wilgenstraat, Roeselare
- Canada (22):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Columbian/Fraser Clinical Trials, New Westminster, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Scarborough Health Network- Rougevalley, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Sherbrooke- Grandby site, Granby, Quebec
  - Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Health Institute, Montreal, Quebec
  - Institut Universitarie de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Kelowna Interior Health, Kelowna
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China
- Germany (10):
  - Klinikum Coburg, Coburg, Bavaria
  - Kerckhoff Klinik, Bad Nauheim, Hesse
  - Herzzentrum Leipzig, Leipzig, Leipzig
  - Herz- und Diabeteszentrum NRW Ruhr-Universitat Bochum, Bad Oeynhausen, North Rhine-Westphalia
  - Elektrophysiologie GFO-Kliniken Bonn, Bonn, North Rhine-Westphalia
  - Herzzentrum der Universitat Koln, Cologne, North Rhine-Westphalia
  - Segeberger Liniken, Bad Segeberg, Schleswig-Holstein
  - UKSH Lubeck, Lübeck, Schleswig-Holstein
  - Universitares Herzzentrum Hamburg, Hamburg
  - ASklepios, Hamburg
- Galilee Medical Centre, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verma A, Birnie DH, Jiang C, Heidbuchel H, Hindricks G, Kirchhof P, Healey JS, Wang Y, Dagres N, Deyell MW, Sanders P, Pathak RK, Koopman P, Nuyens D, Novak P, Amit G, Dussault C, Makanjee B, Quinn FR, Jolly U, Iden L, Kuniss M, Sharma M, Ha A, Essebag V, Champagne J, Hill MD, Smith EE, Wells GA; OCEAN Investigators. Antithrombotic Therapy after Successful Catheter Ablation for Atrial Fibrillation. N Engl J Med. 2026 Jan 22;394(4):323-332. doi: 10.1056/NEJMoa2509688. Epub 2025 Nov 8. PMID 41211931